CLINICAL TRIAL: NCT00811746
Title: Hypnotics to Improve Polysomnography Yield: Eszopiclone vs Ramelteon?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Catherine_Sassoon, Staff Physician, Pricipal Investigator, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: #924
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; eszopiclone; ramelteon; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — ramelteon; Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Rozerem (Ramelteon) 8 mg taken orally 30 minutes before a split-night PSG
  Interventions: Drug: Rozerem (Ramelteon)
- 2 (Active Comparator): Lunesta (Eszopiclone) 3 mg taken 30 minutes before the start of split-night PSG
  Interventions: Drug: Lunesta (Eszopiclone)
- 3 (Other): Historical controls (chart review) matched for demographics and comorbidities of the study drug groups.
  Interventions: Other: Historical Controls

INTERVENTIONS:
Drug: Rozerem (Ramelteon) — 8 mg taken orally 30 minutes before a split-night PSG
  Other Names: Ramelteon
  Arms: 1
Drug: Lunesta (Eszopiclone) — 3 mg taken orally 30 minutes before the start of a split-night PSG
  Other Names: Eszopiclone
  Arms: 2
Other: Historical Controls — Chart review matched for demographics and comorbidities of the study drug groups.
  Arms: 3

SUMMARY:
This study is being conducted to determine if eszopiclone is as effective as ramelteon when used as a pre-medication (sleeping pill) in sleep studies performed to diagnose and treat sleep apnea.

DETAILED DESCRIPTION:
Many Veterans suffer from sleep disordered breathing with a high prevalence of undiagnosed obstructive sleep apnea. One test that can be effective in the diagnosis of sleep apnea is the polysomnogram (PSG). Split-night PSG consists of a diagnostic phase in the first half of the night and a continuous positive airway pressure titration (CPAP) in the second half of the night. CPAP is the standard, most effective therapy for obstructive sleep apnea. Due to the unfamiliar sleep environment of the laboratory and instrumentation that must be used (application of electroencephalogram leads), patients are frequently not able to sleep adequately. In these cases, the PSG must be repeated. Oral hypnotic agents are often used as a pre-medication to increase the yield of PSG in an attempt to decrease the need for repeat studies.

Numerous data is available on the effects of premedication with oral short-acting hypnotics on PSG quality and efficacy of CPAP titration. In one study, eszopiclone, a nonbenzodiazepine gaba-receptor agonist short-acting hypnotic, has been shown to improve PSG quality and CPAP titration. Another short-acting hypnotic, ramelteon, was recently approved by FDA but the effects of ramelteon in improving PSG quality and efficacy of CPAP titration are unclear. The advantage of ramelteon over eszopiclone is the lack of drug dependency or abuse potential. This study aims to evaluate the efficacy of ramelteon compared to eszopiclone when administered prior to split-night PSG and CPAP titration.

ELIGIBILITY:
Inclusion Criteria:

* Referred by VA Long Beach Sleep Clinic at their initial evaluation during outpatient consultation for suspect obstructive sleep apnea.

Exclusion Criteria:

* Sleep disorders other than obstructive sleep apnea
* No prior PSG
* Uncontrolled medical condition
* Prior known adverse reaction to eszopiclone or ramelteon
* Liver disfunction
* Current alcohol abuser
* Current illicit drug abuser
* Alcohol consumption 12 hours prior to polysomnography
* Decompensated psychiatric disorders
* Severe dementia
* Concomitant use of benzodiazepines, trazodone, narcotics, barbiturates or other medications with sedative or hypnotic effects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Non-usable and poor quality PSGs and CPAP intolerance | The morning following the PSG

CONTACTS AND LOCATIONS:
Overall Officials: Catherine S. Sassoon, MD, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Lettieri CJ, Quast TN, Eliasson AH, Andrada T. Eszopiclone improves overnight polysomnography and continuous positive airway pressure titration: a prospective, randomized, placebo-controlled trial. Sleep. 2008 Sep;31(9):1310-6. PMID 18788656
- See also: Southern California Institute for Research and Education Website — http://www.scire-lb.org/